CLINICAL TRIAL: NCT05178810
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of FAB122 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study to Investigate the Efficacy and Safety of FAB122 (Daily Oral Edaravone) in Patients With Amyotrophic Lateral Sclerosis
Acronym: ADORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Collaborators: Julius Clinical (Industry); Stichting TRICALS Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAB122-CT-2001
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAB122 (Experimental)
  Interventions: Drug: FAB122
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FAB122 — Daily dose 100 mg
  Arms: FAB122
Drug: Placebo — Daily dose
  Arms: Placebo

SUMMARY:
Multicenter, multinational, double-blind, randomized (2:1), placebo-controlled Phase III study to investigate the efficacy and safety of 100 mg FAB122 once daily as oral formulation in ALS patients.

ELIGIBILITY:
Main Inclusion Criteria:

* Age 18 - 80 years (both inclusive), male or female;
* Diagnosis of definite, probable, probable laboratory supported or possible ALS as based on the El Escorial and the revised Airlie House diagnostic criteria for ALS;
* Onset of first symptoms* no longer than 24 months prior to randomization;

  *Date of onset is the date the patient reported one or more of the following symptoms:
* Muscle weakness in limbs
* Speech/swallowing difficulties
* Respiratory symptoms: dyspnea was noticed
* SVC equal to or more than 70% of the predicted normal value for gender, height and age at screening visit;
* Change in ALSFRS-R score between 0.35 points and 1.5 points per month (both inclusive) in the period from onset of first symptoms to the Screening visit;
* Capable of providing informed consent and complying with trial procedures.

Main Exclusion Criteria:

* Diagnosis of Primary Lateral Sclerosis;
* Diagnosis of Frontotemporal Dementia;
* Diagnosis of other neurodegenerative diseases (e.g. Parkinson disease, Alzheimer disease);
* Diagnosis of polyneuropathy;
* Other causes of neuromuscular weakness;
* Have a significant pulmonary disorder not attributed to ALS and/or require treatment interfering with the evaluation of ALS on respiratory function;
* Use of intravenous (IV) edaravone within 6 months of the screening visit;
* Depend on mechanical ventilation (invasive or non-invasive) or require tracheostomy at Screening;
* Renal impairment as indicated by a creatinine clearance of less than 50 mL/min as calculated by the Cockcroft Gault equation;
* Subject has a history of clinically significant hepatic disease, hepatitis or biliary tract disease, or subject has a positive screening test for HIV, hepatitis B or C;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- University Hospitals Leuven, Leuven, Belgium
- France (7):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Hospitalo-Universitaire La Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Nice, Nice
  - Hôpital de la Salpêtrière, Paris
  - CHRU de Tours, Tours
- Germany (4):
  - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Hannover Medical School, Hanover
  - Universitätsklinikum Ulm, Ulm
- Trinity College Dublin/Beaumont Hospital, Dublin, Ireland
- Italy (7):
  - Azienda Ospedaliera Universitaria Cagliari, Cagliari
  - Centro Clinico NEMO, Milan
  - University of Milan Medical School, Milan
  - University of Torino - Rita Levi Montalcini Department of Neuroscience, Milan
  - Azienda Ospedaliero Universitaria Di Modena, Modena
  - Azienda Ospedaliera Universitaria ( A O U ) dell'Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - University of Padua - Azienda Ospedaliera di Padova, Padua
- UMC Utrecht, Utrecht, Netherlands
- Poland (3):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - Linden Medical Centre, Krakow
  - City Clinic SP. z o. o., Warsaw
- Centro Hospitalar Universitário Lisboa-Norte, Lisbon, Portugal
- Spain (8):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital San Rafael, Madrid
  - Hospital Universitario La Paz-Carlos III, Madrid
  - Hospital Regional Universitario Málaga, Málaga
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
- Karolinska Institutet, Stockholm, Sweden
- United Kingdom (4):
  - King's College London, London
  - Manchester MND care centre, Manchester
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From the 313 randomized participants, 9 patients were excluded from the analysis and 2 were randomized by mistake and not treated. So a total of 302 participants are considered in the analysis.
Period: Overall Study
Arm/Group | FAB122 | Placebo
Started | 205 | 97
Completed | 155 | 71
Not Completed | 50 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAB122 | Placebo | Total
Number analyzed (Participants) | 205 | 97 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.5) | 59.3 (10) | 59.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 35 | 117
  Male | 123 | 62 | 185
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 185 | 90 | 275
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 6 | 24
Region of Enrollment [Number; unit: participants]
  Europe | 205 | 97 | 302

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) Score After 48 Weeks.
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 171 | 76
units on a scale | -11.2 (7.9) | -10.8 (8.4)

2. Secondary Outcome: Combined Assessment of Function and Survival (CAFS) at 48 and 72 Weeks.
Description: The CAFS (Combined assessment of function and survival) combined information on survival time and ALSFRS-R (ALS Functional Rating Scale-Revised) scores. For this endpoint, each subject's outcome was ranked: the worst subject outcomes received the lowest rank numbers such that a higher CAFS score indicates a better outcome.
  CAFS rankings are computed using:
  Survival data: Patients who die earlier are ranked lower than those who survive longer.
  ALSFRS-R scores: For patients with the same survival duration, ranks are determined by their functional decline (change in ALSFRS-R from baseline).
  For this study the range could go from 1 to 302. Better Outcome: Higher CAFS rank, indicating prolonged survival and/or less functional decline.
  Worse Outcome: Lower CAFS rank, indicating shorter survival and/or greater functional decline.
Time Frame: 48 weeks and 72 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- FAB122 72 Weeks; FAB122 48 Weeks: FAB122: Daily dose 100 mg
- Placebo 72 Weeks; Placebo 48 Weeks: Placebo: Daily dose
Arm/Group | FAB122 72 Weeks | Placebo 72 Weeks | FAB122 48 Weeks | Placebo 48 Weeks
Number analyzed (Participants) | 67 | 33 | 205 | 97
score on a scale | 48.7 (29.41) | 54.15 (28.83) | 153.31 (86.2) | 147.68 (92.38)

3. Secondary Outcome: Survival Probability
Description: Results are based on the overall survival over 72 weeks of treatment, the result is the survival probability estimated over 72 weeks.
  Survival probability is calculated considering time to death, tracheostomy or initiation of non-invasive ventilation for more than 20 hours a day for more than 10 consecutive days, over 72 weeks.
Time Frame: 72 weeks
Measure: Number (95% Confidence Interval); unit: Survival probability
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 67 | 33
Survival probability | 0.728 [0.599 to 0.821] | 0.870 [0.688 to 0.949]

4. Secondary Outcome: Change From Baseline in ALSFRS-R Score After 24 and 72* Weeks
Description: as for outcome 1
Time Frame: 24 weeks, 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FAB122 100mg 24 Weeks; FAB122 100mg 72 Weeks: FAB122 100mg Daily
- Placebo 24 Weeks; Placebo 72 Weeks: Placebo 100mg Daily
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 193 | 93 | 43 | 24
units on a scale | -6.0 (5.4) | -5.4 (5.1) | -15.2 (10.5) | -12.6 (8.2)

5. Secondary Outcome: The Slope of the Decrease in ALSFRS-R Score Over Time at 24, 48 and 72* Weeks;
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  For this outcome, measures on the ALSFRS-R were used to determine the slope of the decrease.
Time Frame: 24, 48, 72 weeks
Measure: Mean (Standard Error); unit: units on a scale/week
Groups:
- FAB122 100mg 24 Weeks; FAB122 100mg 48 Weeks; FAB122 100mg 72 Weeks: FAB122: Daily dose 100 mg
- Placebo 24 Weeks; Placebo 48 Weeks; Placebo 72 Weeks: Placebo: Daily dose
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 205 | 97 | 205 | 97 | 67 | 33
units on a scale/week | -0.2981 (0.0182) | -0.2445 (0.265) | -0.2874 (0.0143) | -0.2767 (0.0206) | -0.3003 (0.0223) | -0.2531 (0.0313)

6. Secondary Outcome: Change From Baseline in ALSFRS-R Score on Bulbar Function (Question 1-3 of the ALSFRS-R) After 24, 48 and 72* Weeks;
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  In this outcome, the Bulbar function (as part of ALSFRS-R) is evaluated, it is related to Speech, Salivation and Swallowing. The maximum score on Bulbar function is 12, and the minimum is 0. Higher score better outcome.
Time Frame: 24, 48 and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 193 | 93 | 171 | 76 | 43 | 24
units on a scale | -1.1 (1.7) | -1.2 (1.6) | -2.1 (2.5) | -2.2 (2.8) | -3.1 (3.5) | -2.7 (2.9)

7. Secondary Outcome: Change From Baseline ALS Functional Rating Scale - Revised Score - Fine Motor Function
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  In this outcome, the fine motor function (as part of ALSFRS-R) is evaluated, it is related to Handwriting, Eating and Cutting food, Dressing and hygiene. The maximum score on fine motor function is 12, and the minimum is 0. Higher score better outcome.
Time Frame: 24, 48 and 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 192 | 93 | 171 | 76 | 43 | 24
units on a scale | -2.0 (2.1) | -1.7 (2.0) | -3.8 (2.9) | -3.3 (2.5) | -4.7 (3.1) | -4.2 (3.3)

8. Secondary Outcome: Change From Baseline ALS Functional Rating Scale - Revised Score - Gross Motor Function
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  In this outcome, the gross motor function (as part of ALSFRS-R) is evaluated, it is related to Climbing stairs, Walking, Rising from a chair. The maximum score on gross motor function is 12, and the minimum is 0. Higher score better outcome.
Time Frame: 24, 48, 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 193 | 93 | 171 | 76 | 43 | 24
units on a scale | -2.0 (1.9) | -1.7 (1.8) | -3.4 (2.7) | -3.3 (2.2) | -4.5 (3.1) | -3.8 (2.4)

9. Secondary Outcome: Change From Baseline ALS Functional Rating Scale - Revised Score - Respiratory Function
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  In this outcome, the respiratory function (as part of ALSFRS-R) is evaluated, it is related to Dyspnea, Orthopnea, Breathing insufficiency. The maximum score on respiratory function is 12, and the minimum is 0. Higher score better outcome.
Time Frame: 24, 48, 72 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 193 | 93 | 171 | 76 | 43 | 24
units on a scale | -0.9 (2.2) | -0.8 (2.1) | -1.9 (3.2) | -2.0 (3.3) | -2.8 (4.2) | -2.0 (2.8)

10. Secondary Outcome: Time to a 3, 6, 9 and 12 Points Change or Death From Baseline in ALSFRS-R Score Over 72* Weeks;
Description: Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
  For this outcome, the time a 3, 6, 9 and 12 points change or death from baseline in ALSFRS-R.
Time Frame: 72 weeks (+/-1 week visit window)
Population: The first 100 patients in the study were planned to complete a 72 weeks follow up. This analysis is done over this population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 67 | 33
days
  Time to 3 points change or death from baseline in ALSFRS-R score | 85 [56 to 169] | 114 [84 to 169]
  Time to 6 points change or death from baseline in ALSFRS-R score | 194 [113 to 286] | 226 [142 to 315]
  Time to 9 points change or death from baseline in ALSFRS-R score | 308 [189 to 504] | 334 [197 to 510]
  Time to 12 points change or death from baseline in ALSFRS-R score | 351 [223 to 511] | 438 [250 to 508]

11. Secondary Outcome: Change in Clinical Staging (King's Staging System and MiToS) Over 72 Weeks
Description: The King's staging system is a simple clinical staging system, which defines 4 stages of ALS. The 1st 3 stages are defined by functional involvement of a region: bulbar, upper limbs, and lower limbs. The number of regions involved gives the stage. Stage 4 is reached if swallowing (4A) or respiratory (4B) difficulty is severe enough to require intervention.
  The outcome of this measure shows the number of patients which staging decline of 1 point or more or No decline.
Time Frame: 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 39 | 24
Participants
  Decline >= 1 | 22 | 12
  No decline | 17 | 12

12. Secondary Outcome: Overall Survival: Proportion of Subjects Alive (Survival Rate) After 24, 48 and 72* Weeks;
Time Frame: 24, 48 and 72* weeks;
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 205 | 97 | 205 | 97 | 67 | 33
proportion of participants | 0.980 [0.947 to 0.992] | 0.990 [0.928 to 0.999] | 0.933 [0.888 to 0.961] | 0.933 [0.857 to 0.970] | 0.791 [0.667 to 0.873] | 0.870 [0.688 to 0.949]

13. Secondary Outcome: Proportion of Subjects Alive and no Tracheostomy, or no Initiation of Non-invasive Ventilation for More Than 20 Hours a Day for More Than 10 Consecutive Days After 24, 48 and 72* Weeks
Time Frame: 24, 48 and 72* weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 205 | 97 | 205 | 97 | 67 | 33
proportion of participants | 0.970 [0.935 to 0.986] | 0.990 [0.928 to 0.999] | 0.903 [0.853 to 0.937] | 0.890 [0.804 to 0.939] | 0.728 [0.599 to 0.821] | 0.870 [0.688 to 0.949]

14. Secondary Outcome: Change From Baseline in Slow Vital Capacity (SVC, Liters) at 24, 48 and 72* Weeks;
Time Frame: 24, 48 and 72* weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 170 | 86 | 129 | 59 | 33 | 20
liters | -0.4 (0.5) | -0.5 (0.7) | -0.7 (0.7) | -0.7 (0.7) | -1 (1) | -1 (0.7)

15. Secondary Outcome: Change From Baseline in the Overall Mega Score for the Hand-held Dynamometer (HHD) at 24, 48 and 72* Weeks.
Description: HHD is a procedure for quantitative strength testing performed in the upper and lower extremities bilaterally. The overall mega score are derived as z-scores of average muscle HHD assessments, percent changes from Baseline are used to derive individual muscle scores.
  Muscle strength is expressed as the percent change from baseline: (post-baselinevalue-baselinevalue)/baselinevalue×100(post-baseline value - baseline value) / baseline value \times 100(post-baselinevalue-baselinevalue)/baselinevalue×100. If the baseline value is zero, the data is considered missing.
  The HDD mega-score averages strength across four muscle locations. It is calculated by averaging the non-missing transformed values. Maximum muscle strength is then standardized using a z-score, based on data from a healthy population.
  Z-score of 0 represents the healthy population mean. Negative z-score value means worse outcome.
Time Frame: 24, 48 and 72* weeks
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 135 | 62 | 109 | 49 | 19 | 16
Z-Score | -0.4 (0.7) | -0.4 (0.6) | -0.7 (1.1) | -0.8 (0.9) | -1.2 (1.2) | -1.4 (0.8)

16. Secondary Outcome: Change From Baseline in the Total Score on the ALS Assessment Questionnaire-40-Item (ALSAQ-40) Form at 24, 48 and 72* Weeks;
Description: ALS Assessment Questionnaire-40-Item. The ALSAQ-40 is specifically used to measure the subjective wellbeing of patients with ALS. There are 40 items/questions in the long form, the ALSAQ-40, with 5 discrete scales: physical mobility (10 items), activities of daily living and independence (10 items), eating and drinking (3 items), communication (7 items), and emotional reactions (10 items). Range is from 0 to 100 scale, where 0 indicates the best quality of life and 100 the worst.
Time Frame: 24, 48 and 72* weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 176 | 83 | 155 | 67 | 40 | 23
units on a scale | 11.2 (12.8) | 8.9 (12.3) | 22.7 (16.8) | 19.9 (17.5) | 27.1 (18.4) | 22.5 (19.5)

17. Secondary Outcome: Change From Baseline in EuroQoL - 5 Dimensions-5 Levels (EQ-5D-5L) Questionnaire Score 24, 48 and 72* Weeks.
Description: European Quality of Life 5 levels and 5 dimensions is a generic questionnaire of health-related quality of life.
  5 Domains: Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression.
  Scale range is from 0 to 100, being 0 the worst and 100 the best.
Time Frame: 24, 48 and 72* weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 205 | 97 | 205 | 97 | 67 | 33
units on a scale
  Anxiety/Depression - Level 1 | 82 (40) | 39 (40.2) | 57 (27.8) | 29 (29.9) | 12 (5.9) | 7 (7.2)
  Anxiety/Depression - Level 2 | 53 (25.9) | 20 (20.6) | 52 (25.4) | 15 (15.5) | 12 (5.9) | 7 (7.2)
  Anxiety/Depression - Level 3 | 39 (19) | 26 (26.8) | 38 (18.5) | 21 (21.6) | 11 (5.4) | 6 (6.2)
  Anxiety/Depression - Level 4 | 12 (5.9) | 3 (3.1) | 12 (5.9) | 4 (4.1) | 6 (2.9) | 4 (4.1)
  Anxiety/Depression - Level 5 | 0 (0) | 0 (0) | 3 (1.5) | 0 (0) | 0 (0) | 0 (0)
  Pain/Discomfort - Level 1 | 66 (32.2) | 33 (34) | 57 (27.8) | 27 (27.8) | 13 (6.3) | 8 (8.2)
  Pain/Discomfort - Level 2 | 61 (29.8) | 26 (26.8) | 47 (22.9) | 19 (19.6) | 10 (4.9) | 8 (8.2)
  Pain/Discomfort - Level 3 | 48 (23.4) | 22 (22.7) | 39 (19) | 19 (19.6) | 12 (5.9) | 6 (6.2)
  Pain/Discomfort - Level 4 | 9 (4.4) | 7 (7.2) | 14 (6.8) | 4 (4.1) | 6 (2.9) | 1 (1)
  Pain/Discomfort - Level 5 | 2 (1) | 0 (0) | 5 (2.4) | 0 (0) | 0 (0) | 1 (1)
  Usual Activities - Level 1 | 21 (10.2) | 10 (10.3) | 10 (4.9) | 4 (4.1) | 1 (0.5) | 1 (1)
  Usual Activities - Level 2 | 35 (17.1) | 8 (8.2) | 22 (10.7) | 4 (4.1) | 4 (2) | 2 (2.1)
  Usual Activities - Level 3 | 50 (24.4) | 31 (32) | 30 (14.6) | 22 (22.7) | 5 (2.4) | 5 (5.2)
  Usual Activities - Level 4 | 41 (20) | 22 (22.7) | 42 (20.5) | 22 (22.7) | 13 (6.3) | 5 (5.2)
  Usual Activities - Level 5 | 40 (19.5) | 16 (16.5) | 57 (27.8) | 17 (17.5) | 18 (8.8) | 11 (11.3)
  Self-care - Level 1 | 36 (17.6) | 11 (11.3) | 16 (7.8) | 5 (5.2) | 3 (1.5) | 1 (1)
  Self-care - Level 2 | 34 (16.6) | 17 (17.5) | 25 (12.2) | 6 (6.2) | 3 (1.5) | 2 (2.1)
  Self-care - Level 3 | 42 (20.5) | 29 (29.9) | 26 (12.7) | 19 (19.6) | 5 (2.4) | 2 (2.1)
  Self-care - Level 4 | 24 (11.7) | 11 (11.3) | 26 (12.7) | 15 (15.5) | 6 (2.9) | 5 (5.2)
  Self-care - Level 5 | 51 (24.9) | 20 (20.6) | 69 (33.7) | 24 (24.7) | 24 (11.7) | 14 (14.4)
  Mobility - Level 1 | 29 (14.1) | 17 (17.5) | 16 (7.8) | 9 (9.3) | 3 (1.5) | 5 (5.2)
  Mobility - Level 2 | 35 (17.1) | 13 (13.4) | 21 (10.2) | 6 (6.2) | 3 (1.5) | 1 (1)
  Mobility - Level 3 | 43 (21) | 19 (19.6) | 29 (14.1) | 14 (14.4) | 6 (2.9) | 2 (2.1)
  Mobility - Level 4 | 49 (23.9) | 27 (27.8) | 49 (23.9) | 21 (21.6) | 14 (6.8) | 7 (7.2)
  Mobility - Level 5 | 31 (15.1) | 12 (12.4) | 47 (22.9) | 19 (19.6) | 15 (7.3) | 9 (9.3)

18. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score at 24, 48 and 72* Weeks.
Description: The Health-Related Quality of Life (HR-QoL) is a questionnaire using a Visual Analog Scale (VAS) ranging from 0 (bad) to 100 (very good).
Time Frame: 24, 48 and 72* weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 182 | 85 | 160 | 67 | 41 | 23
units on a scale | -10.2 (19.4) | -7.2 (23.6) | -15.7 (20.2) | -15.6 (24.9) | -25.1 (21.3) | -15.1 (22.3)

19. Secondary Outcome: Proportion of Subjects With a Change of ≥8, ≥4, and ≥9 for ALS Specific, ALS Non-Specific, and ECAS (Edinburgh Cognitive and Behavioural ALS Screen) Total Score;
Description: The ECAS (Edinburgh Cognitive and behavioural ALS Screen) is a brief multidomain assessment originally designed for people with ALS.
  Total Score Range: 0 to 136 points. Higher scores indicate better cognitive function.
  For ALS-Specific (Assesses cognitive domains most often affected in ALS) Score Range: 0 to 100 points. Higher scores indicate better cognitive function.
  And ALS Non-Specific (Evaluates broader cognitive abilities unrelated to ALS pathology) Score Range: 0 to 36 points. Higher scores indicate better cognitive function.
Time Frame: 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FAB122 100mg 24 Weeks | Placebo 24 Weeks | FAB122 100mg 48 Weeks | Placebo 48 Weeks | FAB122 100mg 72 Weeks | Placebo 72 Weeks
Number analyzed (Participants) | 179 | 88 | 147 | 62 | 35 | 22
Participants
  ALS Specific - Change <8 | 154 | 69 | 128 | 45 | 31 | 18
  ALS Specific - Change >=8 | 25 | 19 | 19 | 17 | 4 | 4
  ALS non-Specific - Change <4 | 153 | 67 | 112 | 46 | 29 | 15
  ALS non-Specific - Change >=4 | 26 | 21 | 35 | 16 | 6 | 7
  ECAS Total Score - Change <9 | 152 | 70 | 121 | 44 | 29 | 19
  ECAS Total Score - Change >=9 | 27 | 18 | 26 | 18 | 6 | 3

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | FAB122 | Placebo
All-Cause Mortality (participants affected / at risk) | 20/205 | 7/97
Serious Adverse Events (participants affected / at risk) | 62/205 | 28/97
Other Adverse Events (participants affected / at risk) | 180/205 | 82/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAB122 (N=205) | Placebo (N=97)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 9 (9)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 6 (7) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Death (General disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femural neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Brain death (General disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Weight decrease (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Utherine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAB122 (N=205) | Placebo (N=97)
COVID-19 (Infections and infestations) | 37 (38) | 14 (14)
Nasopharygitis (Infections and infestations) | 20 (29) | 6 (6)
Urinary tract infection (Infections and infestations) | 15 (18) | 6 (10)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 5 (6)
Constipation (Gastrointestinal disorders) | 25 (25) | 12 (12)
Dysphagia (Gastrointestinal disorders) | 20 (20) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 40 (65) | 27 (52)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 31 (35) | 14 (15)
Nerve conduction studies abnormal (Investigations) | 19 (19) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (20) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 6 (6)
Headache (Nervous system disorders) | 13 (13) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT05178810/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT05178810/SAP_001.pdf